CLINICAL TRIAL: NCT01526031
Title: Randomized Controlled Double Blind Study of Bee Venom Therapy on Adhesive Capsulitis of the Shoulder
Brief Title: Bee Venom Acupuncture for the Treatment of Frozen Shoulder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyunghee University Medical Center (Other)
Collaborators: Kyung Hee University Hospital at Gangdong (Other)
Responsible Party: Principal Investigator, Yonghyeon Baek, Assisstant Professor, Kyunghee University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KHNMC-OH-IRB 2009-013
Record Dates: First submitted 2012-02-01; First posted 2012-02-03 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Frozen Shoulder
Keywords: frozen shoulder; bee venom acupuncture
MeSH Terms: conditions — Bursitis | interventions — Bee Venoms; Acupuncture Therapy; Saline Solution; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- BV1 (Experimental): 1:10,000 bee venom (BV) acupuncture plus physiotherapy
  Interventions: Procedure: 1:10,000 bee venom (BV) acupuncture; Procedure: physiotherapy
- BV2 (Experimental): 1:30,000 bee venom (BV) acupuncture plus physiotherapy
  Interventions: Procedure: 1:30,000 bee venom (BV) acupuncture; Procedure: physiotherapy
- NS (Placebo Comparator): Normal saline injection plus physiotherapy
  Interventions: Procedure: normal saline injection; Procedure: physiotherapy

INTERVENTIONS:
Procedure: 1:10,000 bee venom (BV) acupuncture — after skin test for hypersensitivity to bee venom (0.05ml of 1:30,000 bee venom, SC at LI11)
  * 1st visit : SC 0.4ml of 1:10,000 BV at 4 points (0.1ml for each points)
  * 2nd visit : SC 0.6ml of 1:10,000 BV at 6 points (0.1ml for each points)
  * 3rd visit : SC 0.8ml of 1:10,000 BV at 8 points (0.1ml for each points)
  * 4th to 16th visit : SC 1.0ml of 1:10,000 BV at 10 points (0.1ml for each points)
  Arms: BV1
Procedure: 1:30,000 bee venom (BV) acupuncture — after skin test for hypersensitivity to bee venom (0.05ml of 1:30,000 bee venom, SC at LI11)
  * 1st visit : SC 0.4ml of 1:30,000 BV at 4 points (0.1ml for each points)
  * 2nd visit : SC 0.6ml of 1:30,000 BV at 6 points (0.1ml for each points)
  * 3rd visit : SC 0.8ml of 1:30,000 BV at 8 points (0.1ml for each points)
  * 4th to 16th visit : SC 1.0ml of 1:30,000 BV at 10 points (0.1ml for each points)
  Arms: BV2
Procedure: normal saline injection — after skin test for hypersensitivity to bee venom (0.05ml of 1:30,000 bee venom, SC at LI11)
  * 1st visit : SC 0.4ml of normal saline at 4 points (0.1ml for each points)
  * 2nd visit : SC 0.6ml of normal saline at 6 points (0.1ml for each points)
  * 3rd visit : SC 0.8ml of normal saline at 8 points (0.1ml for each points)
  * 4th to 16th visit : SC 1.0ml of normal saline at 10 points (0.1ml for each points)
  Arms: NS
Procedure: physiotherapy — Physiotherapy treatment will be provided at each visit after bee venom or saline injection.
  * transcutaneous electrical nerve stimulation (TENS) for 15 minutes
  * transcutaneous infrared thermotherapy (TDP) for 15 minutes
  * manual physical therapy for 15 minutes
  * simple home exercise program

SUMMARY:
The purpose of this study is to evaluate the effectiveness of combined bee venom acupuncture (BVA) and physiotherapy (PT) on frozen shoulder, and whether if the effect of BVA is dose effective.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of frozen shoulder by orthopedist
* Must have shoulder pain of more than VAS 5 over 1 month and under 12 months
* Marked limitation of active and/or passive motion range in one shoulder

Exclusion Criteria:

* history of major shoulder injury or surgery
* other musculoskeletal pain
* cervical neuropathy, paralysis, neurological disorder
* hypersensitivity reactions by bee venom skin test
* renal or hepatic disorders, hematologic diseases, cancer, mental disorders, inflammatory or infectious disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2010-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
the Shoulder Pain and Disability Index (SPADI) | Changes from baseline in SPADI at 2, 4, 8, 12 weeks

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) for pain intensity | Changes from baseline in VAS at 2, 4, 8, 12 weeks
passive Range of Motion (pROM) | Changes from baseline in pROM at 2, 4, 8, 12 weeks
  The 4 motions (abduction, forward flexion, extension, and external rotation) will be checked.

CONTACTS AND LOCATIONS:
Overall Officials: Yonghyeon Baek, OMD, Ph.D, Principal Investigator — Kyung Hee University Hospital at Gangdong; Byung-Kwan Seo, OMD, Ph.D, Study Director — Kyung Hee University Hospital at Gangdong
Locations (1):
- Arthritis & Rheumatism Center, Kyung Hee University Hospital at Gangdong, Seoul, South Korea